CLINICAL TRIAL: NCT00631774
Title: An Open Label, Randomized, and Parallel Study to Evaluate the Postprandial Metabolic Response After 24-Week Use of Glucerna SR in Obese Asian Subjects With Type 2 Diabetes
Brief Title: A Study to Evaluate the Postprandial Metabolic Response After Use of Glucerna SR in Obese Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, vghtpe user, Attending physician, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GSR Version 2
Record Dates: First submitted 2008-03-02; First posted 2008-03-10 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: type 2 diabetes; meal replacement; postprandial response; Glucerna SR
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Glucerna

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): a meal replacement program with Glucerna SR on top of the exchange-diet plan
  Interventions: Dietary Supplement: Glucerna SR
- 2 (Active Comparator): an caloric-matched exchange-diet plan only.
  Interventions: Dietary Supplement: Glucerna SR

INTERVENTIONS:
Dietary Supplement: Glucerna SR — Each randomized subject in the meal replacement group will receive Glucerna SR to replace one meal (breakfast) and one pre-sleep snack for 24 weeks. The subjects in the group with exchange-diet plan only will receive a meal plan like they have in the lead-in period.
  Other Names: exchange-diet plan

SUMMARY:
This is a phase 4, 24-week, randomized, parallel, open-label study of a meal replacement program with Glucerna SR in obese Asian participants with type 2 diabetes. The duration of each subject's participation will be approximately 28 weeks, including a lead-in period of 2 weeks and a 2-week post-treatment telephone follow-up. A sufficient number of Asian subjects with type 2 diabetes who have a BMI 18 between 25-40 kg/m2 and meet all the inclusion criteria and none of the exclusion criteria will be entered into the study to randomize approximately 60 subjects. Approximately 60 participants will be randomized to receive either (1) a meal replacement program with Glucerna SR on top of the Exchange-diet plan (EDP) or (2) an caloric-matched EDP only. The primary objective of this study is to evaluate the effect of a diet program including Glucerna SR as a meal replacement on postprandial glucose response after using Glucerna SR for 24 weeks in obese Asian subjects with type 2 diabetes

DETAILED DESCRIPTION:
A sufficient number of Asian subjects (expected to be approximately 90) with type 2 diabetes who have a BMI 18 between 25-40 kg/m2 and meet all the inclusion criteria and none of the exclusion criteria will be entered into the study to randomize approximately 60 subjects. The eligible obese subjects with type 2 diabetes will be entered into a 2-week lead-in period with EDP after individual diet/lifestyle consultation to implement nutrition therapy into their existing diabetes management. The diet recommendations of the EDP at the lead-in period will be based on the nutrition recommendations from the ADA including carbohydrate and monounsaturated fat together provided 60-70 % of energy intake, reduced intakes of saturated fat (< 10 % of total calories) and cholesterol (< 300 mg/day) and protein intake around 15-20 % of total daily energy.

Approximately 60 participants will be randomized at Week 0 (Visit 3) in a 1:1 ratio to receive either (1) a meal replacement program with Glucerna SR on top of the EDP or (2) an caloric-matched EDP only. The participants will receive an educational program of diet, exercise, and behavioral strategies at randomization. Each randomized subject in the meal replacement group will receive Glucerna SR to replace one meal (breakfast) and one pre-sleep snack for 24 weeks. The subjects in the group with EDP only will receive a meal plan like they have in the lead-in period. All study subjects will be placed on a diet plan with 500 ~ 800 kcal/day less than their estimated daily maintenance energy requirement and receive an individualized exercise prescription to facilitate an optimal diabetes management. The participants will visit the clinics at 4-week intervals for 24 weeks after randomization to evaluate the efficacy and the safety parameters. The participants will receive two different meal tests at both the baseline and the end of the study. The macronutrient composition in the meal test protocol 1 is a 480 Kcal Glucerna SR breakfast with 50 % CHO, 20 % protein, and 30 % fat. The test meal protocol 2 is a 480 Kcal sandwich breakfast with 63 % CHO, 20 % protein, and 17 % fat. The primary efficacy variable will be the change from baseline in incremental area under curve (∆AUC) of glucose response after a Glucerna-SR test meal between the two groups.

A telephone follow-up will be performed 2 weeks after the study to evaluate any condition related to the study.

ELIGIBILITY:
Inclusion Criteria:

* Asians
* Diagnosed type 2 diabetes
* BMI between 25 and 40 kgm2
* Aged between 20 and 75 years old
* Current HbA1c between 6.0 and 8.5 percents
* Men and non-pregnant women. If woman, subject is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile, or is of childbearing potential and practicing one of the following methods of birth control-condoms, sponge, foams, jellies, diaphragm or intrauterine device or on contraceptives for the 3-month period prior to Screening-a vasectomized partner-total abstinence from sexual intercourse. If woman, the results of a urine pregnancy test performed at Screening are negative. If woman, subject is not breast-feeding
* Subject is able and willing to replace breakfast and one snack before bed with Glucerna SR
* Subject has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board or Independent Ethics Committee, prior to undertaking any study-specific procedures

Exclusion Criteria:

* History or evidence of type 1 diabetes
* Screening fasting glucose greater than 240 mgdL
* Treatment with insulin, alpha-glucosidase inhibitor, incretin mimetics, or DPP-IV inhibitors in the past 8 weeks
* History of severe hypoglycemia in the past 12 weeks
* History of severe diabetes complications e.g. amputation, blindness, diabetic coma
* Stated history of severe gastroparesis
* Stated significant cardiovascular event e.g., myocardial infarction, stroke within 6 weeks prior to study entry; or stated history of congestive heart failure
* Current use of glucocorticoid steroids with the exception of topical use.
* History of renal insufficiency serum creatinine greater than 1.4 mgdL for women and greater than 1.5 for men
* Subjects with the following laboratory values: hemoglobin less than 10 gdL, WBC less than 3000mL, platelet less than 100,000mL, ALT greater than 3x ULN, total bilirubin greater than 2x ULN
* Stated current severe hepatic disease
* History or evidence of alcoholism or drug abuse
* History or evidence of hyperthyroidism or hypothyroidism
* History of malignancy within the last 5 years
* Consumption of any investigational drug within 30 days prior to enrollment.
* Taking any herbals or dietary supplements during the past 8 weeks that could profoundly affect appetite, weight or glucose metabolism
* Voluntary or involuntary weight loss of greater than 7 percents body weight in past 8 week
* History of major eating disorders, such as anorexia nervosa or bulimia nervosa
* Allergy to Glucerna SR or its content
* History of mental incapacity or language barriers that may preclude adequate understanding or cooperation in the study
* Current or concomitant illness that would interfere with the subject's ability to perform the study or that would confound the study results

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the effect of a diet program including Glucerna SR as a meal replacement on postprandial glucose response after using Glucerna SR for 24 weeks in obese Asian subjects with type 2 diabetes | 24 weeks

SECONDARY OUTCOMES:
evaluate the efficacy and safety of a meal replacement program with Glucerna SR vs. an EDP based on the nutrition therapy recommendations from the ADA on anthropometric measurements, lipid profile, meal-related metabolic changes and quality of life | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Low-Tone Ho, MD, Study Chair — Taipei Veterans eneral Hospital; Chii-Min Hwu, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan